CLINICAL TRIAL: NCT00061516
Title: Safety and Efficacy Study of BETAXON 0.5% and AZOPT 1.0% in Pediatric Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-00-17
Record Dates: First submitted 2003-05-28; First posted 2003-05-30 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — brinzolamide

ARMS (2):
- Brinzolamide suspension, 1% (Experimental): Dosed twice daily for 12 weeks
  Interventions: Drug: AZOPT (brinzolamide)
- Levobetaxolol suspension, 0.5% (Experimental): Dosed twice daily for 12 weeks
  Interventions: Drug: BETAXON (levobetaxolol HCl)

INTERVENTIONS:
Drug: BETAXON (levobetaxolol HCl) — levobetaxolol suspension, 0.5%
  Arms: Levobetaxolol suspension, 0.5%
Drug: AZOPT (brinzolamide) — brinzolamide suspension, 1%
  Arms: Brinzolamide suspension, 1%

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of both BETAXON and AZOPT in pediatric patients. Patients will dose with study drug at 8 am and 8 pm daily for twelve weeks. Patients will have vision tested, slit lamp exam, blood pressure and pulse checks at each visit. Patients will have a dilated fundus exam and corneal measurements taken at first and last visit.

ELIGIBILITY:
INCLUSION:

* Children 5 years old and younger
* require treatment for glaucoma or ocular hypertension
* vision is 20/80 or better
* cup-to-disc ratio of 0.8 or less

EXCLUSION:

* do not have abnormal fixation
* IOP greater than 36 mm Hg
* significant retinal disease
* penetrating keratoplasty
* severe ocular pathology
* optic atrophy
* eye surgery in the past 30 days
* cardiovascular abnormalities
* hypersensitivity to beta blockers, carbonic anhydrase inhibitors or sulfa drugs

Ages: 1 Week to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2003-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline IOP | Up to Week 12

REFERENCES:
- [Result] Whitson JT, Roarty JD, Vijaya L, Robin AL, Gross RD, Landry TA, Dickerson JE, Scheib SA, Scott H, Hua SY, Woodside AM, Bergamini MV; Brinzolamide Pediatric Study Group. Efficacy of brinzolamide and levobetaxolol in pediatric glaucomas: a randomized clinical trial. J AAPOS. 2008 Jun;12(3):239-246.e3. doi: 10.1016/j.jaapos.2007.11.004. Epub 2008 Mar 4. PMID 18289898